CLINICAL TRIAL: NCT03757065
Title: A Cross-Sectional Study of Cell Surface Marker Expression in Participants With Autoimmune or Inflammatory Diseases
Brief Title: Cell Surface Marker Expression in Autoimmune Diseases
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALPN000-001
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Systemic Lupus Erythematosus; Sjogren's Syndrome; Multiple Sclerosis; Systemic Sclerosis; Crohn's Disease; Ulcerative Colitis; Inflammatory Myositis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Multiple Sclerosis; Scleroderma, Systemic; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Systemic Lupus Erythematosus
- Sjogren's Syndrome
- Multiple Sclerosis
- Systemic Sclerosis
- Crohn's Disease
- Ulcerative Colitis
- Inflammatory Myositis

SUMMARY:
This study is designed to explore the expression of cell-surface markers in the following seven disease areas: (a) systemic lupus erythematosus, (b) Sjogren's syndrome, (c) multiple sclerosis, (d) systemic sclerosis, (e) Crohn's disease, (f) ulcerative colitis and (g) inflammatory myositis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 19 years of age or older.
2. Participant or legal surrogate able and willing to provide written, informed consent.
3. Participant is, or has been undergoing care for one of the specified diseases in a participating centre with a confirmed clinical diagnosis of the specified disease.
4. Participant has or will provide the relevant peripheral blood (required) and normal practice tissue specimens (if available).
5. Participant has one of the following target auto-immune or inflammatory diseases diagnosed according to local clinical practice guidelines:

   1. Crohn's Disease
   2. Inflammatory myositis
   3. Multiple sclerosis
   4. Sjogren's syndrome
   5. Systemic lupus erythematosus
   6. Systemic sclerosis
   7. Ulcerative colitis

Exclusion Criteria:

1. Participants receiving investigational therapy within 30 days or 5 half-lives, whichever is longer, prior to enrolment.
2. Participants suffering from any additional disease that may interfere with the biomarker signals as per the investigator's discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with systemic lupus erythematosus, Sjogren's syndrome, systemic sclerosis, multiple sclerosis, Crohn's disease, ulcerative colitis, or inflammatory myositis.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
CD28 Expression | At enrollment
  Percentage of CD28+ T cells in peripheral blood
ICOS Expression | At enrollment
  Percentage of ICOS+ T cells in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hillson, MD, Study Director — Alpine Immune Sciences
Locations (2):
- Canada (2):
  - GI Research Institute, Vancouver, British Columbia
  - Mary Pack Arthritis Center, Vancouver